CLINICAL TRIAL: NCT00702312
Title: A Multi-method Study of a Low-salt Dietary Approach to Control Blood Pressure in the Bangladeshi Chronic Kidney Disease Population.
Brief Title: A Bengali Dietary Salt Study to Control Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: St. Bartholomew's Hospital (Other)
Responsible Party: Ione Ashurst, Barts and The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/Q0605/13
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Study group that will attend low-salt educational community programme
  Interventions: Behavioral: Low-salt educational programme; Behavioral: Low-salt Bangladeshi educational programme
- Control group (No Intervention): Subjects in this arm will have routine medical and dietetic treatment for low-salt reduction.

INTERVENTIONS:
Behavioral: Low-salt educational programme — Subjects will attend a health promotion cooking programme and receive written tailored low-salt Bengali educational tool. This tool has been developed specifically for this population group from Phase 1 and 2 study.
  Other Names: Low-salt health education
  Arms: Study group
Behavioral: Low-salt Bangladeshi educational programme — A multi-component low-salt educational programme tailored to the Bangladeshi kidney disease patients delivered in the community.
  Other Names: Intervention group
  Arms: Study group
Behavioral: Low-salt Bangladeshi educational programme — A multi-component Low-salt educational programme tailored to the Bangladeshi kidney disease patients residents in Tower Hamlets delivered over 5 months.
  Other Names: Intervention group/ Educational group / Low-salt group
  Arms: Study group

SUMMARY:
The aim of this study is to assess the benefits of using low-salt and healthy eating educational programme, designed specifically for Bangladeshi kidney patients, compared to the usual diet advice given by the clinic dietitians.

DETAILED DESCRIPTION:
We conducted an exploratory study initially to learn about the East London Bangladeshi (ELB) kidney patients salt intake. Furthermore, we assessed their educational needs to inform the development and implementation of an educational programme to reduce dietary salt intake in line with the Department of Health recommendations for a good blood pressure control. The educational programme will be tested in a randomized controlled trial. We are interested in salt because studies have shown that salt is one of the causes of high blood pressure. Scientific studies have also shown that the longer a person has high blood pressure the more the damage to the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Adult Bengali kidney disease hypertensive patients

Exclusion Criteria:

* Non-hypertensive Bengali patients and those on dialysis therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reduction in blood pressure | Six months

SECONDARY OUTCOMES:
Reduction in dietary salt intake | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ione Ashurst, BSc, MSc, Principal Investigator — Barts and The London NHS Trust
Locations (1):
- The Royal London Hospital, London, United Kingdom

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] de Brito-Ashurst I, Perry L, Sanders TA, Thomas JE, Dobbie H, Varagunam M, Yaqoob MM. The role of salt intake and salt sensitivity in the management of hypertension in South Asian people with chronic kidney disease: a randomised controlled trial. Heart. 2013 Sep;99(17):1256-60. doi: 10.1136/heartjnl-2013-303688. Epub 2013 Jun 13. PMID 23766446